CLINICAL TRIAL: NCT02062684
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2/3 Study to Evaluate the Efficacy and Safety of Blisibimod Administration in Subjects With IgA Nephropathy
Brief Title: BRIGHT-SC: Blisibimod Response in IgA Nephropathy Following At-Home Treatment by Subcutaneous Administration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-IGN3321
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: IgA Nephropathy
Keywords: IgAN; IgA Nephropathy; A-623; Blisibimod; Kidney Disease; Persistent proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blisibimod (Experimental): Blisibimod administered subcutaneously
  Interventions: Drug: Blisibimod
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blisibimod
  Arms: Blisibimod
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of subcutaneous blisibimod administration in addition to standard therapy in patients with biopsy proven IgA Nephropathy with persistent proteinuria of between 1-6 g/day.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age, inclusive
* Biopsy-proven IgA nephropathy
* Receiving stable, clinically-optimized ACEI and/or ARB
* Proteinuria ≥ 1g/24hr but ≤ 6g/24hr at 2 consecutive time points

Exclusion Criteria:

* Clinical or histologic evidence of non-IgA-related glomerulonephritis
* IgA nephropathy with greater than 50% glomerulosclerosis or cortical scarring
* Meets eGFR criteria
* History of treatment with oral or parenteral corticosteroids within 3 months or immunosuppressants within 6 months
* Malignancy within past 5 years
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C
* Liver disease
* Neutropenia
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections
* History of active tuberculosis or a history of tuberculosis infection
* Pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving reduction in proteinuria from baseline | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in serum immunoglobulins IgA, IgG and IgM | 24 weeks
Percent reduction from baseline in plasma cells and B-cell subsets | 24 weeks
Percent change from baseline in complement C3 and C4 | 24 weeks
Proportion of subjects progressing to End Stage Renal Disease | Approximately 104 weeks
Proportion of subjects achieving reduction in proteinuria from baseline | Approximately 104 weeks
Numbers of subjects requiring the addition of corticosteroid or other therapy | 24 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- Czechia (2):
  - Investigator Site 852, Olomouc
  - Investigator 851, Prague
- Investigator Site 905, Düsseldorf, Germany
- Investigator Site 101, Hong Kong, Hong Kong
- Investigator Site 603, Kajang, Malaysia
- Philippines (2):
  - Investigator Site 402, Quezon City
  - Investigator Site 401, Quezon City
- Singapore (2):
  - Investigator Site 202, Singapore
  - Investigator Site 201, Singapore
- South Korea (5):
  - Investigator Site 305, Busan
  - Investigator Site 306, Busan
  - Investigator Site 303, Daejeon
  - Investigator Site 301, Seoul
  - Investigator Site 302, Seoul
- Taiwan (2):
  - Investigator Site 704, Changhua
  - Investigator Site 705, Tainan
- Thailand (4):
  - Investigator Site 504, Bangkok
  - Investigator Site 505, Bangkok
  - Investigator Site 503, Bangkok
  - Investigator Site 501, Chang Mai
- United Kingdom (3):
  - Investigator Site 806, Bradford
  - Investigator Site 801, Leicester
  - Investigator Site 803, London

REFERENCES:
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537